CLINICAL TRIAL: NCT02167529
Title: A Prospective, Multicenter and Observational Trial to Evaluate Evolution of Quality of Life (SF-36) After Total Thyroidectomy.
Brief Title: Quality of Life After Thyroidectomy (ThyrQol)
Acronym: ThyrQol
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC11_0194
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Total Thyroidectomy
Keywords: Quality of life-Thyroidectomy-Morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the evolution of quality of life and voice function with different questionnaires (VIH, SF36) before and after total thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years
* Notice to total thyroidectomy
* Thyroidectomy under cervicotomy or videoscopy
* Existence of a written informed consent of the patient
* Affiliation to a social security
* Possible follow-up for 6 months

Exclusion Criteria:

* Impossibility for the patient to complete the forms
* Impossibility to follow the patient patient with serious disease which impact the quality of life
* Medullary thyroid cancers
* Preoperative examination of vocal cords (if performed) finding a violation of the vocal cords
* Lack of monitoring possible during the 6 months after surgery
* Pregnant women or during lactation
* Minors and adults under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective, non randomized, open, multicenter trial to evaluate quality of life (SF 36) and voice function (VHI questionnaire) before and after totalthyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 890 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the differences in terms of impact on quality of life among patients without sequelae 6 months after thyroidectomy (laryngeal paralysis or hypoparathyroidism) and patients with hypoparathyroidism. (SF36 v1,3, self-administered questionnaire) | Evaluation at 6 months

SECONDARY OUTCOMES:
Evaluation of the impact of post thyroidectomy laryngeal paralysis on the quality of life (SF36 v1,3, self-administered questionnaire) | Evaluation at 2 and 6 months
Evaluation of difficulties voice after total thyroidectomy (with or without laryngeal complication) (VIH questionnaire) | Evaluation at 2 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Mirallié, Pr, Principal Investigator — Nantes University Hospital
Locations (7):
- France (7):
  - Angers University Hospital, Angers
  - CHD La Roche sur Yon, La Roche-sur-Yon
  - Limoges University Hospital, Limoges
  - Lyon University Hospital, Lyon
  - Nancy University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - La Pitié-Salpétrière - AP-HP, Paris